CLINICAL TRIAL: NCT05162677
Title: Prophylactic Mastectomy: Prospective Evaluation of the Correlation Between Skin Flap Thickness, Residual Glandular Tissue and Skin Necrosis by Imaging and Clinical Examination
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Rebecka Wiberg, Resident in plastic surgery, PhD, Umeå University
Other Study IDs: 2021-PrMa-RWiberg
Record Dates: First submitted 2021-10-27; First posted 2021-12-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Prophylactic Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most common form of cancer among women. Five to ten percent of all breast cancers are due to hereditary factors, with pathogenic variants in the breast cancer genes BRCA1/2 accounting for 2-5% of all breast cancer. Women with pathogenic variants in BRAC1/2 and other pathogenic gene mutations leading to an increased risk of breast cancer can undergo prophylactic mastectomy, reducing the risk of breast cancer up to 90%. Among women who have undergone prophylactic mastectomy, 1-1,9% are diagnosed with breast cancer, but little is known about the correlation between residual glandular tissue and skin flap thickness, as well as the oncological risk of residual glandular tissue. Furthermore, there is a balance between how much subcutaneous tissue should be resected to achieve maximal reduction of glandular tissue, while leaving viable skin flaps. In addition, there are established surveillance guidelines for women with pathogenic variants in BRCA1/2 who do not undergo risk-reducing surgery, but no published consensus or guidelines regarding appropriate medical follow-up for those who opt for prophylactic mastectomy. The aim of this study is to investigate the correlation between skin flap thickness, residual glandular tissue and skin flap necrosis following prophylactic mastectomy in women with results from postoperative magnetic resonance tomography, ultrasound and physical examination, as well as evaluate patient satisfaction and quality of life pre- and postoperatively with different questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women that are recommended prophylactic mastectomy at the Department of Plastic Surgery at Umeå University hospital due to hereditary factors that have been investigated by clinical geneticists.
* Age between 18-74 years

Exclusion Criteria:

* Women undergoing mastectomy due to cancer.
* Age < 18 years or > 74 years.

Ages: 18 Years to 74 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All women with elevated risk of developing breast cancer due to hereditary factors that will undergo prophylactic mastectomy at the Department of Plastic Surgery at Umeå University hospital and forfill the inclusion criteria will be invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of residual glandular tissue | Residual glandular tissue will be evaluated 1 year postoperatively
  Residual glandular tissue will be reported as being present or not present through postoperative evaluation with magnetic resonance tomography, ultrasound and mammography. The quadrants of the left and right breast will be examined after which the findings will be documented in pre-printed templates.
Presence of residual glandular tissue | Residual glandular tissue will be evaluated 3 years postoperatively
  Residual glandular tissue will be reported as being present or not present through postoperative evaluation with magnetic resonance tomography, ultrasound and mammography. The quadrants of the left and right breast will be examined after which the findings will be documented in pre-printed templates.
Measurement of skin flap thickness | Skin flap thickness will be evaluated 1 year postoperatively
  The skin flap thickness will be evaluated postoperatively with magnetic resonance tomography, ultrasound and mammography. The quadrants of the left and right breast will be examined after which the findings will be documented in pre-printed templates. The skin flap thickness will be defined as the thickness of the skin (epidermis, dermis, subcutaneous tissue) measured at the examinations rather than the thickness of the skin flaps perioperatively. All measurements will be made in mm.
Measurement of skin flap thickness | Skin flap thickness will be evaluated 3 years postoperatively
  The skin flap thickness will be evaluated postoperatively with magnetic resonance tomography, ultrasound and mammography. The quadrants of the left and right breast will be examined after which the findings will be documented in pre-printed templates. The skin flap thickness will be defined as the thickness of the skin (epidermis, dermis, subcutaneous tissue) measured at the examinations rather than the thickness of the skin flaps perioperatively. All measurements will be made in mm.

SECONDARY OUTCOMES:
Change in evaluation of patient satisfaction | Change in patient satisfaction will be evaluated pre- and postoperatively. The women will receive the questionnaires 1 month preoperatively, 1 year postoperatively and 3 years postoperatively.
  Patient satisfaction will be evaluated pre- and postoperatively with four different validated questionnaires; BREAST-Q, BRECON23, QLQ-C30 and Cancer-worry scale.
Change in evaluation of patient quality of life | Change in patient quality of life will be evaluated pre- and postoperatively. The women will receive the questionnaires 1 month preoperatively, 1 year postoperatively and 3 years postoperatively.
  Patient quality of life will be evaluated pre- and postoperatively with four different validated questionnaires; BREAST-Q, BRECON23, QLQ-C30 and Cancer-worry scale.
Number of participants with acute postoperative complications | Clinical examination will be performed 2-4 weeks postoperatively.
  Postoperative complications will be evaluated postoperatively by clinical examination and documented in pre-printed templates, and pictures will be taken. The complications will include breast related complications (skin flap necrosis, infection, hematoma, seroma and implant loss) and non-breast related complications (deep vein thrombosis, pulmonary embolism).
Number of participants with long term postoperative complications | Clinical examination will be performed 1 year postoperatively.
  Postoperative complications will be evaluated postoperatively by clinical examination and documented in pre-printed templates, and pictures will be taken. The complications will include breast related complications (skin flap necrosis, infection, hematoma, seroma and implant loss) and non-breast related complications (deep vein thrombosis, pulmonary embolism).
Number of participants with long term postoperative complications | Clinical examination will be performed 3 years postoperatively.
  Postoperative complications will be evaluated postoperatively by clinical examination and documented in pre-printed templates, and pictures will be taken. The complications will include breast related complications (skin flap necrosis, infection, hematoma, seroma and implant loss) and non-breast related complications (deep vein thrombosis, pulmonary embolism).

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic Surgery Unit, Umeå University hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The study is currently a single center study but might in the future be expanded to a multicenter study. Furthermore, someone else with a different study question might want to use the cohort later on.

REFERENCES:
- [Background] Wiberg R, Andersson MN, Svensson J, Rosen A, Koch F, Bjorkgren A, Sund M. Prophylactic Mastectomy: Postoperative Skin Flap Thickness Evaluated by MRT, Ultrasound and Clinical Examination. Ann Surg Oncol. 2020 Jul;27(7):2221-2228. doi: 10.1245/s10434-019-08157-2. Epub 2020 Jan 6. PMID 31907748
- [Background] Skoglund MA, Andersson MN, Bjorkgren A, Tolocka E, Sund M, Wiberg R. Inter- and intra-observer agreement on evaluating the presence of residual glandular tissue with magnetic resonance tomography following prophylactic mastectomy. Acta Radiol. 2023 Jan;64(1):67-73. doi: 10.1177/02841851211058929. Epub 2021 Dec 1. PMID 34851154